CLINICAL TRIAL: NCT03988270
Title: Presurgical Arm Exercises Prior to Creation of a Forearm AV Fistula in Hemodialysis (HD) Patients With End-stage Kidney Disease: A Pilot Study
Brief Title: Prefistula Forearm Exercise in Pts Requiring Chronic HD Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00058671
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-06

CONDITIONS: Arterio-venous Fistula; Kidney Failure; Hemodialysis Access Failure
Keywords: Hemodialysis; Fistula; Access Failure; Hemodialysis Fistula Creation
MeSH Terms: conditions — Arteriovenous Fistula; Renal Insufficiency; Fistula | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized study with two arms: Intervention arm with a pre-fistula placement exercise program versus a control arm with no prefistula placement exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participant randomized to an exercise protocol using a hand grip device that is used on a daily basis. Participant will be encouraged to increase the number of repetitions used by the hand grip device during the course of the trial
  Interventions: Other: Exercise
- Control (No Intervention): Participants in the control group will not receive any pre-surgical instructions for exercise in the access arm

INTERVENTIONS:
Other: Exercise — Participant randomized to an exercise protocol using a hand grip device that is used on a daily basis. Participant will be encouraged to increase the number of repetitions used by the hand grip device during the course of the trial
  Arms: Exercise

SUMMARY:
For chronic hemodialysis patients, the creation of a well-functioning arteriovenous (AV) fistula is critical for ensuring that patient receive adequate hemodialysis. Unfortunately, the primary failure rate for AV fistulas after surgery is about 40%, and this percentage has not changed despite a number of trials of pharmaceutical agents and biologic agents. A key to success in the development of a useable AV fistula is an adequate arterial and venous diameter in the access forearm. Although exercise is commonly used to increase vessel diameter after AV fistula placement, Investigators are unaware of published studies that report on the effect of exercise prior to AV fistula placement to assist with the maturation of a newly created AV fistula. In this pilot trial, the Principal Investigator will evaluate the feasibility and possible benefits of pre-surgical exercise on forearm AV fistulas.

DETAILED DESCRIPTION:
The trial is designed to determine if a pre-surgical exercise program will improve the likelihood of a useable forearm AV fistula. In this pilot study, the feasibility of the proposed intervention will be assessed in terms of both patient acceptability and patient outcomes. In addition, results from this feasibility study will be used to help determine power calculations for a full-scale trial.

Patients will be eligible for this pilot clinical trial if scheduled for placement of an elective forearm AV fistula for chronic hemodialysis access. Patients will be randomized using a random number generator to either the intervention or the control group. The intervention group will be instructed in the use of hand grip with built in digital counter. These instructions will include the use of the hand grip on a daily basis with an increasing number of hand grip squeezes to be performed each week up until the time of fistula placement.

Patients in the control group will not receive any pre-surgical instructions for exercise in the access arm. In both groups, patients will be provided with post-surgical instructions on the use of a squeeze ball on a daily basis once the steri-strips from the surgical site have fallen off.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for placement of an elective forearm AV fistula for chronic hemodialysis access.

Exclusion Criteria:

* The presence of joint or musculoskeletal impairments that prevent the patient from using a handgrip device on a daily basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with fistula usable without intervention | Up to 12 weeks after surgical creation of the AV fistula
  Fistula usability will be measured by the use of the AV fistula for two needle cannulation for chronic dialysis sessions within 12 weeks after surgical creation.
Number of participants with fistula usable with intervention | Up to 12 weeks after surgical creation of the AV fistula
  Fistula usability will be measured by the use of the AV fistula for two needle cannulation for chronic dialysis sessions within 12 weeks after surgical creation.
Number of participants with fistula not usable | Up to 12 weeks after surgical creation of the AV fistula
  Fistula usability will be measured by the use of the AV fistula for two needle cannulation for chronic dialysis sessions within 12 weeks after surgical creation.

SECONDARY OUTCOMES:
Mean Number of hand grips per day | Up to 8 weeks after start of the intervention
Mean Number of days hand grips performed | Up to 8 weeks after start of the intervention
Total mean number of hand grip repetitions performed | Up to 8 weeks after start of the intervention
Cephalic Vein Doppler measurement | Up to 8 weeks after start of the intervention
  The diameter of the vessel in centimeters will be measured using a Duplex Doppler.
Basilic Vein Doppler measurement | Up to 8 weeks after start of the intervention
  The diameter of the vessel in centimeters will be measured using a Duplex Doppler.
Median Cubital Doppler measurement | Up to 8 weeks after start of the intervention
  The diameter of the vessel in centimeters will be measured using a Duplex Doppler.
Radial Artery Doppler measurement | Up to 8 weeks after start of the intervention
  The diameter of the vessel in centimeters will be measured using a Duplex Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rocco, MD, MSCE, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03988270/ICF_000.pdf